CLINICAL TRIAL: NCT00544154
Title: Efficacy and Safety of CDP870 400 mg in Combination With Methotrexate Compared to Methotrexate Alone in the Treatment of the Signs and Symptoms of Patients With Rheumatoid Arthritis Who Are Partial Responders to Methotrexate
Brief Title: Efficacy and Safety of CDP870 and Methotrexate Compared to Methotrexate Alone in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C87014
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Arthritis, Rheumatoid
Keywords: CDP870; Certolizumab pegol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CDP870

SUMMARY:
The main purpose of the study was to determine the efficacy of CDP870 in treating RA signs/symptoms in patients who were partial responders to MTX. Other purposes were to show additional efficacy without increased toxicity and the immunogenic response to CDP870 during combined CDP870 and MTX therapy.

ELIGIBILITY:
Inclusion Criteria:

* male/female, 18-75 years old, inclusive
* diagnosis of adult-onset RA
* had active disease
* had received methotrexate
* on a stable dose of folic acid

Exclusion Criteria:

* contraindication for methotrexate or anti-TNF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2002-10; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
American college of Rheumatolofy (ACR)-20 responder rate at Week 24

SECONDARY OUTCOMES:
Safety and tolerability
health outcomes measures
immunogenic profile of CDP870 plus methotrexate
systemic exposure of CDP870

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Choy E, McKenna F, Vencovsky J, Valente R, Goel N, Vanlunen B, Davies O, Stahl HD, Alten R. Certolizumab pegol plus MTX administered every 4 weeks is effective in patients with RA who are partial responders to MTX. Rheumatology (Oxford). 2012 Jul;51(7):1226-34. doi: 10.1093/rheumatology/ker519. Epub 2012 Feb 16. PMID 22344576